CLINICAL TRIAL: NCT03934996
Title: Quality and Behavior of Pelvic Floor in Runner Women
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Stopped PhD project
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Dr. Antonio I Cuesta-Vargas, Principal Researcher of CTS631 University of Malaga, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: corredorasSP
Record Dates: First submitted 2019-04-22; First posted 2019-05-02 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Pelvic Floor Disorders; Sport Injury; Stress Urinary Incontinence
Keywords: pelvic floor; athletes
MeSH Terms: conditions — Pelvic Floor Disorders; Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The researcher will not know who belongs to each group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Assesment Runners (No Intervention): Healthy woman between 25 and 44 years old, not pregnant and running at least 10 km/week.
- Runners with educational training (Experimental): Healthy woman between 25 and 44 years old, not pregnant and running at least 10 km/week with educational training about pelvic floor muscles.
  Interventions: Other: Runners with educational training

INTERVENTIONS:
Other: Runners with educational training — Intervention will consist of an educational talk to know the anatomy and function of the Pelvic Floor Muscles and 20 minutes of both strength and endurance exercises with biofeedback. An exercise protocol will be carried out. The participants will be instruct to contract and maintain maximum force for a mean period of 6 seconds (endurance training) and rest for twice the length of the endurance training time, followed by three fast contractions in a row as strength training. It will be done twice a week, during 12 weeks.
  Pelvic floor assesment: Perineometry, manual palpation, electromyography Trunk and lower limbs electromyography and kinematics
  Arms: Runners with educational training

SUMMARY:
The main objective is to analyze the relationship between the PF muscles and the other variables along the different tasks of daily life and during the race.

DETAILED DESCRIPTION:
Introduction: Women are more likely to suffer injuries in the Pelvic Floor (PF) and Urinary Incontinence (UI) because of their anatomical characteristics. Their participation in the sports field has been more active recently. There are studies that correlate the race with presenting weakness of the SP muscles and Stress Urinary Incontinence (SUI), so the race is considers as a risk factor for these affectations. However, there are few studies of real-time measurements during running. Some runners may even present SUI during daily activities (ADL). The UI is not only a physical problem but also affects the social, emotional, psychological, sexual and professional level and may even lower their self-esteem or renounce the physical activity.

Objectives: The purpose of this study is to perform measurements of different variables in real time while running and in their ADL. The main objective is to analyze the relationship between the PF muscles and the other variables along the different tasks of daily life and during the race. The secondary objectives are to differentiate these neuromuscular, physiological and biomechanical responses of PF and abdominal girdle (AG) according to the type of stroke, duration, intensity and distance. And compare results between both group (interventional group and no interventional group).

Material and method: Randomized clinical trial will be performed with 59 female runners aged 25-44 years. The sample will be divided into two groups randomly. The study will be carried out health center called "Tiro de Pichón" in Málaga.

ELIGIBILITY:
Inclusion Criteria:

* Healthy woman between 25 and 44 years old.
* Women not pregnant.
* Women who run at least 10 km / week.
* In case of having children, it has to be 12 months after childbirth, having had the first postpartum menstruation and having left breastfeeding.

Exclusion Criteria:

* Women Pregnant or suspected of it.
* Postpartum less than one year.
* Having the period during the exploration for the classification in groups or during the day of the measurements.
* Present operation in the urogenital region as well as any visceral or spinal operation.
* Urinary tract and/or vaginal infections.
* Vaginal lesions; anorectal lesions or bleeding.
* Women with gynecological bleeding; urethral obstruction; fistulas; malformations (ectopic ureter, etc); genital prolapse.
* Women with pain in Pelvic Floor or lower limbs or back.
* Pain during the race.
* Allergy to silver, nickel and/or latex.

Ages: 25 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 0 (Actual)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change %MVC | Prior and after intervention, an average of 12 weeks
  Change % of Maximun voluntary contraction
Change of Base Tone of Pelvic Floor Muscles (EMG) | baseline, prior and after intervention, an average of 12 weeks
  Electromyography of base tone of Pelvic Floor Muscles
Change of step length | Prior and after intervention, an average of 12 weeks
  Metres of the step length. It will measure with two cinematic shimmers wich will be placed on both tibias.
Change of cadence | Prior and after intervention, an average of 12 weeks
  steps/secons. It will measure with two cinematic shimmers wich will be placed on both tibias.It will measure with a cinematic shimmer wich will be placed on both tibias.
Change of ground reaction force | Prior and after intervention, an average of 12 weeks
  Newton of the ground reaction force. It will measure with two cinematic shimmers wich will be placed on both tibias.
Change of acceleration | Prior and after intervention, an average of 12 weeks
  Change of Acceleration (m/s2 axes X, Y, Z). It will measure with a EXG shimmer wich will be placed on the sternun.
Change of displacement | Prior and after intervention, an average of 12 weeks
  metres of displacement. It will measure with two cinematic shimmers wich will be placed on both tibias.
Change of accumulated fatigue | Prior and after intervention, an average of 12 weeks
  Using Lactate Pro 2. Mmol/Litres
Change of heart rate | Prior and after intervention, an average 12 weeks
  Heart Rate
Perineometry of MCV | baseline, prior and after intervention, an average of 12 weeks
  perineometry of MCV using PFX
Intravaginal manual palpation | baseline, prior and after intervention, an average of 12 weeks
  manual testing of the levator ani muscles using scale of Daniels
Change of electromyography of Pelvic Floor Muscles | Prior and after intervention, an average of 12 weeks
  Change of electromyography of Pelvic Floor Muscles

SECONDARY OUTCOMES:
Change Pelvic floor functional capacity | Prior and after intervention, an average of 12 weeks
  Difference between Perineometry of MCV and Base Tone of Pelvic Floor Muscles (EMG)
Quality of life score | Prior and after intervention, an average of 12 weeks
  Using SF-12 health survey scoring demonstration. It provides a profile of the state of health and is one of the most commonly used generic scales in the evaluation of clinical outcomes. It is a self-administered instrument of 12 items from the 8 dimensions of the SF-36: Physical Function (2), Social Function (1), Physical Role (2), Emotional Role (2), Mental Health (2), Vitality (1) ), Corporal Pain (1), General Health (1). For each of the 8 dimensions, the items are coded, aggregated and transformed into a scale that ranges from 0 (the worst state of health for that dimension) to 100 (the best state of health). Validated by Ware J Jr, Kosinki M, Meller SD. and the Spanish version by Vilagut et al., 2008, who obtained an internal consistency coefficient of about 0.9 for Sf-36 and lower light for SF-12. The Cronbach alpha coefficients of the summary components of the SF-12 exceeded the proposed minimum of 0.7 for group comparisons.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Malaga, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hagovska M, Svihra J, Bukova A, Horbacz A, Drackova D, Svihrova V, Kraus L. Prevalence of Urinary Incontinence in Females Performing High-Impact Exercises. Int J Sports Med. 2017 Mar;38(3):210-216. doi: 10.1055/s-0042-123045. Epub 2017 Feb 17. PMID 28212587
- [Background] Chevalier F, Fernandez-Lao C, Cuesta-Vargas AI. Normal reference values of strength in pelvic floor muscle of women: a descriptive and inferential study. BMC Womens Health. 2014 Nov 25;14:143. doi: 10.1186/s12905-014-0143-4. PMID 25420756
- [Background] Leitner M, Moser H, Eichelberger P, Kuhn A, Radlinger L. Evaluation of pelvic floor muscle activity during running in continent and incontinent women: An exploratory study. Neurourol Urodyn. 2017 Aug;36(6):1570-1576. doi: 10.1002/nau.23151. Epub 2016 Oct 29. PMID 27794169
- [Background] Luginbuehl H, Naeff R, Zahnd A, Baeyens JP, Kuhn A, Radlinger L. Pelvic floor muscle electromyography during different running speeds: an exploratory and reliability study. Arch Gynecol Obstet. 2016 Jan;293(1):117-124. doi: 10.1007/s00404-015-3816-9. Epub 2015 Jul 21. PMID 26193953
- [Background] Goldstick O, Constantini N. Urinary incontinence in physically active women and female athletes. Br J Sports Med. 2014 Feb;48(4):296-8. doi: 10.1136/bjsports-2012-091880. Epub 2013 May 18. PMID 23687004
- [Background] Bo K. Urinary incontinence, pelvic floor dysfunction, exercise and sport. Sports Med. 2004;34(7):451-64. doi: 10.2165/00007256-200434070-00004. PMID 15233598
- [Background] Carvalhais A, Da Roza T, Vilela S, Jorge RN, Bo K. Association Between Physical Activity Level and Pelvic Floor Muscle Variables in Women. Int J Sports Med. 2018 Dec;39(13):995-1000. doi: 10.1055/a-0596-7531. Epub 2018 Oct 16. PMID 30326528